CLINICAL TRIAL: NCT06427057
Title: A Prospective, Open Label, Dual Cohort Study of Cadonilimab（AK104）Combined With Standard Treatment for Function Preservation in Urinary System Tumors
Brief Title: A Study of Cadonilimab（AK104）Combined With Standard Treatment for Function Preservation in Urinary System Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Liu Huang, Clinical Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20240519
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Urinary System Tumor
Keywords: UC，RCC，immunotherapy, neoadjuvant
MeSH Terms: conditions — Urologic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC (Experimental): Patients will receive AK104 (10mg/kg ,Q3W，intravenously) plus standard regimen （gemcitabine or albumin paclitaxel) neoadjuvant treatment with no more than 6 cycles.
  Interventions: Drug: Cadonilimab plus chemotherapy
- RCC (Experimental): Patients will receive AK104 (10mg/kg ,Q3W，intravenously) plus standard regimen （TKI，e.g. sunitinib, pezopanib) neoadjuvant treatment with no more than 6 cycles.
  Interventions: Drug: Cadonilimab plus TKI

INTERVENTIONS:
Drug: Cadonilimab plus chemotherapy — AK104 (10mg/kg ,Q3W，intravenously) plus chemotherapy（e.g. gemcitabine or albumin paclitaxel，dosage based on guidelines or instructions）
  Arms: UC
Drug: Cadonilimab plus TKI — Patients will receive AK104 (10mg/kg ,Q3W，intravenously) plus TKI（e.g. sunitinib, pezopanib，dosage based on guidelines or instructions)
  Arms: RCC

SUMMARY:
This is an open label, dual cohort ,phase II study to explore efficacy and safety of cadonilimab(PD-1/CTLA-4 Bispecific Antibody) combined with standard regimen neoadjuvant treatment in urothelial carcinoma（UC） and renal cell carcinoma（RCC）, with evaluating successful preservation rate of bladder/kidney.

DETAILED DESCRIPTION:
UC and RCC confirmed by histopathology or cytology prior have not received systematic treatment, who had indications for surgical resection and were difficult to preserve organ function after surgery or were partially resection but the patients have a strong desire to preserve organ function. This study enrolled 20 cases in each cohort of UC and RCC，pts received neoadjuvant treatment containing cadonilimab for no more than 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary agreement to provide written informed consent.
* Male or female, Age ≥ 18 years.
* Predicted survival ≥ 12 weeks.
* Histologically confirmed diagnosis of urothelial carcinoma（UC） and renal cell carcinoma（RCC）.
* Prior no antitumor systematic treatment .
* Have clinically non-metastatic high risk urothelial carcinoma (cT2-T4a, N0-3, M0) .
* High risk renal cell carcinoma (≥ T2Nx or TanyN+)，include subjects with only Oligotransfer.
* Willing to undergo surgical resection and were difficult to preserve organ function after surgery or were partially resection but the patients have a strong desire to preserve organ function.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment.
* Male and female participants are eligible to participate if they agree to the contraception use as per study protocol.
* Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

* Has received other antitumor therapy before planned start of trial treatment.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive, or HIVAb positive.
* Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
* NYHA Class III heart failure.
* Suffering from active infection requiring systemic treatment.
* Uncontrolled hypertension, diabetes, Interstitial lung Disease, or COPD;
* Treated with systemic treatment (e.g. immunomodulators, corticosteroids or immunosuppressants) for the autoimmune disease within 2 years prior to the study treatment.
* History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Pregnancy or lactation.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Bladder/Kidney Preservation rate | Up to approximately 18 Weeks (Time of surgery)
  Evaluating the impact of neoadjuvant therapy on organ preservation function

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 18 Weeks
  percentage of participants with a complete response (CR) or partial response (PR)
Rate of Pathologic Response | Up to approximately 18 Weeks (Time of surgery) ]
  No residual tumor (ypT0N0) and partial response (ypTis-1N0) in surgical specimen.
Overall Survival (OS) | Up to approximately 36 Months
  Overall survival is defined as the time from enrollment to death due to any cause.
Assess Adverse Events | 12 months
  Assess adverse events according to the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Liu Huang, Clinical Professor, Principal Investigator — Tongji Hospital , Wuhan, Hubei Province, China, 430030; Xiao Yu, Clinical Professor, Principal Investigator — Tongji Hospital , Wuhan, Hubei Province, China, 430030